CLINICAL TRIAL: NCT01945476
Title: Effect of Midazolam Premedication Before Induction on the Functional Recovery After General Anesthesia in the Patients Undergoing Breast Surgery Due to Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2013-0444
Record Dates: First submitted 2013-09-04; First posted 2013-09-18 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Breast Cancer
Keywords: midazolam; premedication; functional recovery; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- midazolam (Experimental): midazolam group
  Interventions: Drug: midazolam premedication
- normal saline (Active Comparator): control group
  Interventions: Drug: midazolam premedication

INTERVENTIONS:
Drug: midazolam premedication — On the day when patients are scheduled for operation, one researcher will use a computer to randomly select and allocate patients. By randomization, patients will be divided into two groups, receiving an injection of either 0.02 mg/kg of midazolam(midazolam group) or saline (control group). The researcher who randomly allocated patients will prepare the medicines but not just medicine. Investigators must mix it with normal saline to obtain a total volume of 5 mL and label two of them all "prepared medicine," never letting the doctors and subjects know which is midazolam and which is saline.
  Use the QoR-40 survey form to investigate the functional recovery of the patient. This survey will be administered before the operation and on the first and second days after the operation; it will be administered three times in total.

SUMMARY:
Normally, higher levels of preoperational stress or anxiety affect behavior and recovery after the operation. Moreover, patients undergoing mastectomy are usually young women, and this demographic is known to experience higher levels of stress and anxiety than any other. Anesthetizing patients involves more than just anesthesia in operation; it also includes all of the preoperative treatments for optimizing a patient's condition and promoting quick postoperative recovery. Pharmacological premedication for anxiolysis or amnesia before anesthesia has been a common means of sedation that many studies have investigated. However, such studies have focused on alleviating patients' anxiety and on how far patients can obey induction for sedation; there has been no research on post-operational prognoses, the ultimate purpose of reducing anxiety.

The well-known effect of pharmacological premedication is to reduce the capacity of the anesthetic. However, it is not confirmed whether this effect leads to better recovery after anesthesia, as this question has not been researched. Furthermore, recently some have argued strongly that premedication actually prolongs recovery and that it does not need to be applied to every patient. Recently, therefore, the use of pharmacological premedication has been left to the discretion of institutes or doctors in many cases.

Among types of premedication, midazolam belongs to the class of short-acting benzodiazepines and is frequently used, as it induces meaningful anterograde amnesia and causes fewer aftereffects such as respiratory problems. In addition, its effects have already been demonstrated. However, research on the improvement of functional health after anesthesia-i.e., patients' quick return to normal life-is still poor and needs to be advanced.

When measuring the degree of recovery, recent studies tend to focus on measuring how quickly patients are able to return to normal life rather than the recovery of specific symptoms. To this end, the most widely used method is the Quality of Recovery 40 (QoR-40) survey. It has a total of 40 items, which are classified into five categories: emotional state, physical comfort, psychological support, physical independence, and pain. Questions are answered using a 5-point scale, with 1 being worst and 5 being best. It takes 6.3 minutes on average to complete, and its test-retest reliability, internal consistency, and split-half coefficient have led it to be recognized as the most effective survey method. Moreover, it has been used in many studies investigating how the type of operation, method of anesthesia, additional medication, and gender affect anesthesia and the operation. Its validity for such research has been verified.

Therefore, investigators can investigate the degree of postoperational functional recovery through the QoR-40 by comparing cases in which an operation is performed with or without midazolam.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 20 and 65 years who are scheduled to undergo mastectomy because of breast cancer, who are classified as 1-2 according to the American Society of Anesthesiologists (ASA) physical status classification, and who use Korean as their mother tongue will be chosen as participants after obtaining informed consent from them; some may be excluded from participation according to certain criteria.

Exclusion Criteria:

* Patients who recently have been taking medicine that can affect the CNS, such as sedatives and sleeping pills
* people who drink more than one bottle of alcohol every day
* patients with prior experience of anesthesia or operation
* people with a BMI of 30 or higher
* pregnant women
* patients who are known to be allergic to propofol
* patients whose breasts are going to be dissected and then immediately re-constructed using their own body tissue.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The QoR-40 administered 24 hours after the operation is the primary endpoint of this research. | 24 hours after the operation
  The researchers unaware of patients' group assignment will come to visit each patient before the operation and on the first and second days after the operation and administer the QoR-40 survey. They will evaluate the quality of recovery after general anesthesia by considering the global score (200 points in total) of QoR-40 surveys, which is obtained by summing the subtotal scores for emotional status, physical comfort, psychological support, physical independence, and pain. The QoR-40 administered 24 hours after the operation is the primary endpoint of this research. If there is a difference of 10 points or more between those two groups, we will consider that there is a significant difference between them.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain MedicineSeverance Hospital, Yonsei University Health System, Seoul, South Korea